CLINICAL TRIAL: NCT01474902
Title: A Randomized Controlled Trial of Enoxaparin in Children With Asymptomatic Venous Thrombosis After Pediatric Cardiac Surgery
Brief Title: Enoxaparin in Children With Asymptomatic Venous Thrombosis After Pediatric Cardiac Surgery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian McCrindle, Staff Cardiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000022022
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Asymptotic Venous Thrombosis
Keywords: pediatric; asymptotic venous thrombosis; Enoxaparin; pediatric cardiac surgery
MeSH Terms: interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): The initial enoxaparin dose will be: 1.75 mg/kg/dose SC q12h for patients ≤ 2 months old or
  1 mg/kg/dose SC q12h for patients > 2 months old
  Adjust the dose of enoxaparin according to the following monogram. Depending on the Enoxaparin Anti-factor Xa level achieved, successive actions are indicated, including whether to hold the next scheduled dose, whether any dose change is indicated and when the next anti-factor Xa level should be drawn.
  Interventions: Drug: Enoxaparin
- No-treatment (No Intervention)

INTERVENTIONS:
Drug: Enoxaparin — Lovenox- Enoxaparin; Sanofi-Aventis Canada Inc.
  Arms: Treatment group

SUMMARY:
The CATCH-enoxaparin trial is the natural continuation of the CATCH study. It will capitalize on the fact that patients enrolled in the CATCH study will be specifically screened for asymptomatic thromboembolism (TEs) in order to answer important clinical questions.

The investigators propose a randomized controlled trial to address whether, among pediatric patients with congenital heart defects (CHD) recovering from cardiovascular surgery and diagnosed with an asymptomatic venous TE, the use of enoxaparin results in a net therapeutic benefit?

DETAILED DESCRIPTION:
Primary Aim: To address whether, among pediatric patients with congenital heart defects (CHD) recovering from cardiovascular surgery and diagnosed with an asymptomatic venous TE, the use of enoxaparin results in a net therapeutic benefit. We hypothesize that enoxaparin dosed as per age-appropriate algorithms is associated with an increased rate of clot resolution and decreased rate of clot progression/long-term complications in children with CHD and asymptomatic venous TE. Benefits from clot resolution will outweigh the risks associated with the use of enoxaparin resulting in a net therapeutic benefit in favour of enoxaparin use in this context.

Secondary aims of this study are to:

1. To compare the rate of conversion from asymptomatic to symptomatic TE and/or thromboembolic events between treated and untreated patients. Hypothesis: the use of enoxaparin will significantly reduce the rate of conversion from asymptomatic to symptomatic TE.
2. To compare the rate of objective clot progression (or regression) by serial imaging with ultrasound and echocardiography between treated and untreated patients. Hypothesis: the use of enoxaparin will significantly increase the rate of clot regression.
3. To identify factors associated with: TE conversion from asymptomatic to symptomatic, clot resolution and post-thrombotic syndrome in both treated and untreated patients separately. Hypothesis: older children with a more mature coagulation system and those with TEs in superficial vessels (rather than deep/systemic vessels) will have a lower frequency of TE complications.
4. To establish the rate of bleeding complications (both minor and major) for patients on enoxaparin. Hypothesis: we expect major bleeding complications to be present in 2-3% of treated patients and minor bleeding complications to be frequent.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients with a cardiac defect (acquired or congenital)
2. Recent cardiac surgery (during current hospital admission)3) Presence of a venous clot confirmed by appropriate diagnostic imaging methods associated with either ≥ 25% blood vessel occlusion (clot diameter/vessel diameter) OR is ≥ 3mm in absolute diameter
3. Enrollment in the Heart Centre Biobank Registry
4. Enrollment in the CATCH main study

Exclusion Criteria:

1. Clots associated with any of the following symptoms: swelling, edema, discoloration or high temperature of the affected territory.
2. Clots in a vascular segment/location (arterial clots, intracardiac clots) or with a degree of vessel occlusion which obligatory warrants treatment
3. Prosthetic heart valve
4. Active or previous cancer history
5. Known congenital coagulopathy or thrombophilic disorder
6. Liver failure (AST, ALT or % bilirubin 2x normal)
7. Need for anticoagulation for treatment or prophylaxis for other reasons (e.g. BT shunt, recent thrombosis requiring anticoagulation)
8. Previous documented residual clot within the same vascular territory affected by current asymptomatic clot
9. Increased bleeding risk reflected by severe thrombocytopenia (platelet count <30,000/ml) and/or coagulopathy (INR >4.0 or aPTT >120s)
10. Active bleeding or major bleeding <10 days ago (not surgery related)
11. Previous neurosurgery <14 days ago
12. Uncontrolled severe hypertension (>95th percentile for age)
13. Previous proven diagnosis of heparin-induced-thrombocytopenia (HIT) <100 days ago
14. Absolute contraindication to heparin/LMWH (e.g. severe heparin allergy)
15. Pregnancy or breastfeeding
16. No planned follow-up at The Hospital for Sick Children

While most patients will be identified as part of the CATCH study during the pre-discharge full-body vascular ultrasound, some patients who are not enrolled in CATCH will also be identified if an asymptomatic clot is identified during a clinically indicated radiological study. For those patients who are not already enrolled in the CATCH study and the Heart Centre Biobank Registry, they will be approached and consent will be obtained for those studies prior to enrolment in the CATCH-enoxaparin study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Net therapeutic benefit of enoxaparin | Events recording from baseline to 18 months post-surgery
  Defined as the between group difference in proportion of patients with negative outcomes (percent clot conversion to symptomatic + percent major bleeding complications)

SECONDARY OUTCOMES:
Rate of objective clot size progression (or regression) | Up to 18 months post-surgery
  This will be determined by serial imaging with ultrasound and frequency of complete clot resolution at the end of the treatment
Frequency and Risk Factors for conversion from asymptomatic to symptomatic thromboembolism | Up to 18months post-surgery
  Defined as the appearance of any of the following symptoms: swelling, edema, discoloration or high temperature of the affected territory
Frequency of and risk factors for post-thrombotic syndrome | 18 months after surgery
  Clinical manifestations include varicose veins, edema, skin hyperpigmentation and skin ulcers
Frequency of and risk factors for bleeding complications | Up to 18months
  Minor complications and major episodes defined as cerebral, abdominal, retroperitoneal or pulmonary hemorrhage or any bleeding complications requiring blood transfusions
Neurodevelopment and health re-lated quality of life | 18 months post-surgery
  Age appropriate PedsQL® generic module and parent report and Child Health Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Brian W McCrindle, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada